CLINICAL TRIAL: NCT04068220
Title: Intraoperative Continuous Flash Visual Evoked Potentials Monitoring During Minimally Invasive Endoscopic Skull Base Surgery, a Novel Approach to Improve Patient Outcome
Brief Title: Intraoperative Continuous Flash Visual Evoked Potentials Monitoring During Endoscopic Skull Base Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fahad AlKherayf (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Fahad AlKherayf, Associate Scientist, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190533 - 01H
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Chiasmal; Lesion; Prechiasmal; Lesion
Keywords: chiasmal, prechiasmal, lesion, endoscopic skull base surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative FVEPs monitoring (Other): adult patients admitted to TOH - Civic Campus, for chiasmal or pre-chiasmal lesions undergoing a first time minimally invasive endoscopic skull base surgery.
  Interventions: Other: intraoperative FVEPs monitoring

INTERVENTIONS:
Other: intraoperative FVEPs monitoring — During the surgery, a pair of goggles (similar to the swimming goggles) will be placed on patient's closed eyes. The goggles equipped with red LEDs will apply no pressure or minimal pressure on patient's closed eyes. Patient's left eye then right eye will be stimulated with flashing red light emitted by the goggles. Two subdermal needle electrodes will be placed under the skin behind patient's ears, and one subdermal needle electrode will be placed under the skin above the bridge of patient's nose. The two electrodes placed behind patient's ears, will record intraoperative flash visual evoked potentials (FVEPs) resulted from red light stimulation of patient's visual pathway through the eyes and the electrode above the bridge of the nose will record, at the same time, the activity of each eye's retina.

SUMMARY:
Skull base surgeries performed in areas involving the visual pathway are associated with varying levels of postoperative visual dysfunction. The goal of intraoperative FVEP monitoring is to detect and prevent intraoperative visual pathway injury.

DETAILED DESCRIPTION:
Skull base surgeries performed in areas involving the visual pathway are associated with varying levels of postoperative visual dysfunction. For instance, surgical resection of suprasellar meningiomas has been shown to worsen visual function in 14 - 28% of patients and surgical resection of craniopharyngiomas worsen visual function in 3 - 11.5% of patients. Manipulation of the optic nerve and interference with the microvasculature during surgical dissection is thought to be responsible for the visual loss.

Through intraoperative monitoring and prompt identification of flash visual evoked potentials (FVEPs) deterioration, corrective surgical measures could be undertaken to improve or stabilize postoperative visual dysfunction. Furthermore, intraoperative FVEPs monitoring may influence surgical decision-making thus contributing to predict and prevent postoperative visual dysfunction as well as allowing more total resection of a tumour when the monitoring is stable.

This study's aim is to determine if intraoperative continuous FVEPs monitoring can predict and prevent or minimize possible visual pathway injury that may appear during minimally invasive endoscopic skull base surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult population (18 years and older), admitted to The Ottawa Hospital (TOH)-Civic Campus for a chiasmal or pre-chiasmal lesion, undergoing first time minimally invasive endoscopic skull base surgery
* Patient able to personally sign and date the informed consent document
* Patients will be selected based on the surgeon's determination that:

  1. The visual system will be at risk of iatrogenic injury
  2. The intraoperative FVEPs monitoring could rapidly detect this injury AND
  3. Corrective measures could be taken during surgery to reverse it.

Exclusion Criteria:

* patients having a pre-existent retinal disease, cardiac pacemaker
* contraindication for total intravenous anaesthesia (TIVA)
* unable to complete required pre and post-operative visual assessment or unable to complete their post-operative follow-up visits at TOH-Civic Campus
* anticipated goggle movement related to reflection of the frontal skin flap
* preoperative visual deficits (e.g., profound deficits in visual acuity or dense visual field loss)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine the feasibility of detecting iatrogenic visual pathway injury by using intraoperative monitoring of continuous FVEPs in minimally invasive endoscopic skull base surgery. | 1 year
  This pilot study will evaluate the number of enrolled patients with stable and reliable FVEPs with ERGs, the number of enrolled patients with more than 50% decrease in intraoperative FVEPs N1-P1 amplitude (compared to baseline value) and the number of patients with permanent postoperative visual deficit. In addition, we will use demographic data for descriptive analysis, and obtain preliminary data for power analysis and information on subject recruitment before starting the large clinical trial.

SECONDARY OUTCOMES:
Determine sensitivity and specificity as well as positive and negative predictive value of intraoperative monitoring of continuous FVEPs in minimally invasive endoscopic skull base surgery. | 1 year
  Evaluation of proportions (sensitivity and specificity) and performances (positive and negative predictive values)
Report the adverse events of intraoperative monitoring continuous FVEPs | 1 year
  Determine the number and percentage of each identified adverse event of intraoperative continuous FVEPs monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alkherayf, MD MSc FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - Civic Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Ottawa Hospital website — http://www.ottawahospital.on.ca